CLINICAL TRIAL: NCT01962259
Title: Active Commuting To Improve Well-being and Health in Everyday Life
Acronym: GO-ACTIWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Bente Merete Stallknecht, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACTIWE-1
Record Dates: First submitted 2013-09-25; First posted 2013-10-14 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vigorous intensity LTPA (Experimental): Leisure time physical activity (LTPA): Exercise intensity: 70% of maximal oxygen uptake (VO2 max); Energy expenditure: Females: 1600 kcal/week; Males: 2100 kcal/week
  Interventions: Behavioral: Physical activity
- Moderate intensity LTPA (Experimental): Leisure time physical activity (LTPA): Exercise intensity: 50% VO2 max; Energy expenditure: Females: 1600 kcal/week; Males: 2100 kcal/week
  Interventions: Behavioral: Physical activity
- Active commuting (Experimental): Bicycling to/from work/school/university. No requirements for exercise intensity; Energy expenditure: Females: 1600 kcal/week; Males: 2100 kcal/week; Avg distance per day Females 9-15 km; Males 11-17 km
  Interventions: Behavioral: Physical activity
- Control (No Intervention): Receives no intervention.

INTERVENTIONS:
Behavioral: Physical activity
  Arms: Active commuting; Moderate intensity LTPA; Vigorous intensity LTPA

SUMMARY:
The aim of present randomized controlled trial is to evaluate the health effects of physical activity in transport and leisure time domains of everyday life and to develop durable physical activity regimens, i.e. to go from lifestyle intervention to daily lifestyle routine, in overweight individuals.

Subjects will be randomized to 1 of 4 groups. 1: Vigorous intensity leisure time physical activity, 2: Moderate intensity leisure time activity, 3: Active commuting by bicycle, or 4: a non-intervention control group

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No engagement in habitual structured physical activity
* Body mass index 25-35 kg/m2
* Body fat percentage >32% for women and >25% for men
* Maximum oxygen uptake (VO2max) <40 ml O2/kg/min for women and <45 ml O2/kg/min for men
* Ethnicity: Caucasian

Exclusion Criteria:

* Chronic use of medicine
* Smoking
* Fasting plasma glucose > 6,1 mmol/L
* Blood pressure > 140/90 mm Hg
* Abnormal resting and working ECG
* Parents or siblings with diagnosed type 2 diabetes
* For women: Follicle stimulating hormone (FSH) concentration > 35 milliunits/ml, pregnancy or planning of pregnancy within the coming year

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity (glucose clearance ml/min/kg fat-free mass/nM insulin) | Change from baseline in peripheral insulin sensitivity at 3 months
  Measured using the hyper-insulinemic euglycaemic clamp
Peripheral insulin sensitivity (glucose clearance ml/min/kg fat-free mass/nM insulin) | Change from baseline in peripheral insulin sensitivity at 6 months
  Measured using the hyper-insulinemic euglycaemic clamp
Haemostatic balance | Change from baseline in endogenous thrombin potential at 3 months
  Blood coagulation measured by fasting levels of endogenous thrombin potential (nM x min)
Haemostatic balance | Change from baseline in endogenous thrombin potential at 6 months
  Blood coagulation measured by fasting levels of endogenous thrombin potential (nM x min)

SECONDARY OUTCOMES:
Glycaemic control | Baseline, 3 and 6 months
  Fasting plasma glucose, 1- and 2-hour plasma glucose and glucose area under the curve measured during an oral glucose tolerance test
Central insulin sensitivity | Baseline, 3 and 6 months
  Fasting plasma insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test
Maximal oxygen uptake (ml/O2/kg/min) | Baseline, 3 and 6 months
  Measured using indirect calorimetry and an incremental bicycle protocol
Abdominal fat mass | Baseline, 3 and 6 months
  Visceral intrabdominal and subcutaneous fat mass determined by magnetic resonance imaging
Metabolic syndrome | Baseline, 3 and 6 months
  As measured by high density lipoprotein, triglycerides, waist circumference, blood pressure, mean arterial pressure, fasting glucose and composite metabolic syndrome scores
Haemostatic balance II | Baseline, 3 and 6 months
  1: Coagulation: Fibrinogen, Tissue factor(TF), prothrombin fragment 1+2. 2: Fibrinolysis: Tissue type plasminogen activator(tPA:AG), Plasminogen activator inhibitor type 1(PAI-1:AG). 3: Endothelial cell function: von Willebrand factor(vWF), Tissue factor pathway inhibitor (TFPI). 4: Inflammation: C-Reactive protein.
Health related quality of life and other psycho-social outcomes | Baseline, 3 and 6 months
  Measured using questionaries (SF-36), semi-structured interviews and observations
Anthropometry | Baseline, 3 and 6 months
  Measured using dual x-ray absorptiometry, height, weight, waist and hip circumference, sagittal abdominal height
Sleep habits | Baseline, 3 and 6 months
  Sleep duration and quality measured using accelerometers, logs and questionaires (Pittsburgh sleep quality index and Epworth sleepiness scale)
Skeletal muscle biopsy | Baseline, 3 and 6 months
  Biochemical, proteomics, metabolomics, genomics and morphological analyses
Subcutaneous adipose tissue biopsy | Baseline, 3 and 6 months
  Biochemical, proteomics, metabolomics, genomics and morphological analyses

OTHER OUTCOMES:
Exercise compliance | Baseline, 3 and 6 month
  Adherence to the exercise protocol as measured using heart rate and global positioning system monitors will be assessed and individually adjusted continuously over the course of the exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bente M Stallknecht, MD,PHD,DMSc, Principal Investigator — University of Copenhagen, Department of Biomedical Sciences
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Derived] Kern T, Blond MB, Hansen TH, Rosenkilde M, Quist JS, Gram AS, Ekstrom CT, Hansen T, Stallknecht B. Structured exercise alters the gut microbiota in humans with overweight and obesity-A randomized controlled trial. Int J Obes (Lond). 2020 Jan;44(1):125-135. doi: 10.1038/s41366-019-0440-y. Epub 2019 Aug 29. PMID 31467422
- [Derived] Quist JS, Rosenkilde M, Gram AS, Blond MB, Holm-Petersen D, Hjorth MF, Stallknecht B, Sjodin A. Effects of Exercise Domain and Intensity on Sleep in Women and Men with Overweight and Obesity. J Obes. 2019 Apr 7;2019:2189034. doi: 10.1155/2019/2189034. eCollection 2019. PMID 31089425
- [Derived] Blond MB, Rosenkilde M, Gram AS, Tindborg M, Christensen AN, Quist JS, Stallknecht BM. How does 6 months of active bike commuting or leisure-time exercise affect insulin sensitivity, cardiorespiratory fitness and intra-abdominal fat? A randomised controlled trial in individuals with overweight and obesity. Br J Sports Med. 2019 Sep;53(18):1183-1192. doi: 10.1136/bjsports-2018-100036. Epub 2019 Mar 16. PMID 30878970
- [Derived] Quist JS, Rosenkilde M, Petersen MB, Gram AS, Sjodin A, Stallknecht B. Effects of active commuting and leisure-time exercise on fat loss in women and men with overweight and obesity: a randomized controlled trial. Int J Obes (Lond). 2018 Mar;42(3):469-478. doi: 10.1038/ijo.2017.253. Epub 2017 Oct 10. PMID 28993707
- [Derived] Gram AS, Bladbjerg EM, Quist JS, Petersen MB, Rosenkilde M, Stallknecht B. Anti-inflammatory effects of active commuting and leisure time exercise in overweight and obese women and men: A randomized controlled trial. Atherosclerosis. 2017 Oct;265:318-324. doi: 10.1016/j.atherosclerosis.2017.06.923. Epub 2017 Jun 28. PMID 28679486